CLINICAL TRIAL: NCT01858454
Title: A Randomized Controlled Trial of Hand-assisted Laparoscopic Myomectomy Versus Abdominal Myomectomy: Surgical Outcomes and Patient Satisfactions
Brief Title: Hand-assisted Laparoscopic Surgery (HALS) for Myomectomy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study enrollment is not enough
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KNC13-012
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Uterine Myomas
MeSH Terms: interventions — Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HALS for myomectomy (Experimental): Hand-assisted laparoscopic surgery for myomectomy
  Interventions: Procedure: HALS
- Open myomectomy (Active Comparator): Open surgery for myomectomy
  Interventions: Procedure: Open surgery

INTERVENTIONS:
Procedure: HALS — In HALS, a trocar of 5-mm calipers was inserted through the umbilicus. Next, suprapubic transverse skin incision of 3-4cm in length was made and a wound retractor (Alexis; Applied Medical, Rancho Santa Margarita, CA) was inserted through the suprapubic opening.
  Arms: HALS for myomectomy
Procedure: Open surgery — In open surgery, the patient was placed in the supine position and the operation was carried out in a standard manner as described elsewhere [Luciano AA. Myomectomy. Clin Obstet Gynecol 2009;52:362-71.].
  Arms: Open myomectomy

SUMMARY:
The aim of this study was to evaluate the feasibility and usefulness of Hand-assisted laparoscopic surgery (HALS) for myomectomy, and compare it with the open approach in myomectomy.

DETAILED DESCRIPTION:
Uterine myomas are the most common benign tumor of the female genital tract and the leading indication for hysterectomy. Despite the fact that laparoscopic myomectomy is becoming increasingly popular, laparoscopic myomectomy remains underutilized because of inherit limitations. The limitations include technical challenges such as dissection of the myoma from its bed using the correct plane or multilayer closure of the myoma bed and the concern about the strength of the suturing and the subsequent risk of uterine rupture. As a result, laparoscopic myomectomy is currently performed only by expert surgeons.

Hand-assisted laparoscopic surgery (HALS) is a unique surgical approach that may overcome the limitations of pure laparoscopic surgery. HALS is not only less invasive than open surgery but also causes less technical challenges than laparoscopic surgery based on its manual nature and ability to use retractors. In gynecologic field, HALS has also been employed in ovarian cancers and large ovarian tumors.

In theory, HALS seems appropriate procedure, similar to the open approach, for patients with multiple or huge myomas. To date, no report has evaluated the feasibility and usefulness of HALS compared with open surgery (OS).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were as follows: women who had myoma-related symptoms such as menorrhagia, pelvic pressure/pain, or infertility; women who were not pregnant at the time of presentation (i.e., negative for urine pregnancy test or last menstrual period within the last 4 weeks); and women who were appropriated medical status for laparoscopic surgery (American Society of Anesthesiologists Physical Status classification 1 or 2).

Exclusion Criteria:

Exclusion criteria included any other uterine or adnexal abnormalities (e.g., abnormal endometrial thickness, and suspected ovarian or uterine malignancy), any sign of genital infection, presence of submucosal or pedunculated myoma as a dominant myoma, treatment of gonadotropin-releasing hormone (GnRH) agonist 2 months before surgery, or an inability to understand and provide written informed consent.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction about surgery | 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD, Principal Investigator — CHA Gangnam Medical Center, CHA university, Seoul, Republic of Korea
Locations (1):
- CHA Gangnam Medical Center, Seoul, South Korea